CLINICAL TRIAL: NCT01075321
Title: A Phase I/II Clinical Trial of the mTor Inhibitor RAD001 (Everolimus) in Combination With Lenalidomide (Revlimid) for Patients With Relapsed or Refractory Lymphoid Malignancy
Brief Title: Everolimus and Lenalidomide in Treating Patients With Relapsed or Refractory Non-Hodgkin or Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0981; NCI-2010-00235 (Registry Identifier: NCI-CTRP); 09-003801 (Other: Mayo Clinic IRB); RV-NHL-HL-PI-0466 (Other: Celgene Protocol); CRAD001NUS113T (Other: Novartis Protocol); MC0981 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Waldenstrom Macroglobulinemia | interventions — Everolimus; Lenalidomide; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry; Microarray Analysis; Gene Expression Profiling; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral everolimus once daily and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: lenalidomide; Other: laboratory biomarker analysis; Genetic: polymorphism analysis; Other: immunohistochemistry staining method; Genetic: microarray analysis; Genetic: fluorescence in situ hybridization

INTERVENTIONS:
Drug: everolimus — Given orally
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Other: laboratory biomarker analysis — Correlative studies
Genetic: polymorphism analysis — Correlative studies
Other: immunohistochemistry staining method — Optional correlative studies
  Other Names: immunohistochemistry
Genetic: microarray analysis — Optional correlative studies
  Other Names: gene expression profiling
Genetic: fluorescence in situ hybridization — Optional correlative studies
  Other Names: fluorescence in situ hybridization (FISH)

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Giving everolimus together with lenalidomide may be an effective treatment for lymphoma.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving everolimus and lenalidomide together and to see how well they work in treating patients with relapsed or refractory non-Hodgkin or Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.Phase I: To establish the maximum tolerated dose of EVEROLIMUS and lenalidomide in subjects with relapsed/refractory Non-Hodgkin Lymphoma or Hodgkin Lymphoma.

II. Phase II: To assess tumor response to EVEROLIMUS and lenalidomide in subjects with relapsed/refractory Non-Hodgkin Lymphoma or Hodgkin Lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate overall survival, progression-free survival, duration of response, and time to treatment failure of subjects receiving EVEROLIMUS and lenalidomide.

II. To describe the adverse event profile (using CTCAE CTEP Version 4.0) of EVEROLIMUS and lenalidomide.

OUTLINE: Patients receive oral everolimus once daily and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* Histological or cytological confirmation of relapsed or refractory non-Hodgkin lymphoma or Hodgkin lymphoma =< 6 months prior to registration
* The following disease types are eligible: Study 1 - Aggressive lymphomas- Transformed lymphomas; Diffuse large B cell lymphoma; Mantle cell lymphoma; Follicular lymphoma grade III; Precursor B lymphoblastic leukemia/lymphoma; Mediastinal (thymic) large B-cell lymphoma; Burkitt lymphoma/leukemia; Precursor T lymphoblastic leukemia/lymphoma; Primary cutaneous anaplastic large cell lymphoma; and Anaplastic large cell lymphoma-primary systemic type
* Study 2- Indolent lymphomas: Follicular lymphoma, grades 1, 2; Extranodal marginal zone B-cell lymphoma of MALT type; Nodal marginal zone B-cell lymphoma; Splenic marginal zone B-cell lymphoma; Small lymphocytic lymphoma
* Study 3- Uncommon lymphomas: Peripheral T cell lymphoma, unspecified; Anaplastic large cell lymphoma (T and null cell type); Lymphoplasmacytic lymphoma (Waldenstrom Macroglobulinemia); Post transplant lymphoproliferative disorders; Mycosis fungoides/Sezary syndrome; Hodgkin Disease; Primary effusion lymphoma; Adult T-cell leukemia/lymphoma; Extranodal NK/T-cell lymphoma, nasal type; Enteropathy-type T-cell lymphoma; Hepatosplenic T-cell lymphoma; Subcutaneous panniculitis-like T-cell lymphoma; Angioimmunoblastic T-cell lymphoma; Anaplastic large cell lymphoma-primary cutaneous type; and Blastic plasmacytoid dendritic cell neoplasm
* Measurable disease by CT or MRI or PET/CT: Must have at least one lesion that has a single diameter of >= 2 cm or tumor cells in the blood >= 5 x10^9/L (Skin lesions can be used if the area is >= 2 cm in at least one diameter and photographed with a ruler)
* For lymphoplasmacytic lymphoma patients without measurable lymphadenopathy, measurable disease is defined by both of the following criteria: Bone marrow lymphoplasmacytosis with > 10% lymphoplasmacytic cells or aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy and quantitative IgM monoclonal protein > 800 mg/dL
* ANC >= 1200/uL
* Hgb > 9 g/dl
* PLT >= 50,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN the direct bilirubin must be normal
* AST =< 2.5 x ULN or AST =< 5 x ULN if liver involvement
* Creatinine =< 1.5 x ULN
* Creatinine clearance >= 50mL/min (Cockcroft-Gault calculation)
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN (NOTE: Lipid lowering medication is allowed)
* ECOG Performance Status (PS) 0, 1, or 2
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test with a sensitivity of at least 50 IU/ml within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide, during study treatment and for 8 weeks after the last dose of RAD001 (FCBP must also agree to ongoing pregnancy testing)
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy (All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure)
* Provide informed written consent
* Willingness to return to Mayo Clinic enrolling institution for follow-up
* Patient is willing to provide blood samples for research purposes
* Recovered from acute side effects of prior myelosuppressive chemotherapy or biological therapy
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist

Exclusion

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Active other malignancy, excepting non-melanotic skin cancer or carcinoma-in-situ of the cervix (If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer)
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects; Nursing women; Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the study and for 8 weeks after the last dose of study drug (NOTE: If barrier contraceptives are being used, these must be continued throughout the trial by both sexes; hormonal contraceptives are not acceptable as a sole method of contraception)
* Patients who have received prior treatment with both an mTOR inhibitor (sirolimus, temsirolimus, everolimus) and lenalidomide who did not have a response to either when used as single agents
* Patients with a known allergic reaction to thalidomide, RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or their excipients to the point where either agent should not be given again
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Known positive for HIV or infectious hepatitis, type A, B or C
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Prior Allogeneic Stem Cell Transplant
* No chronic treatment with systemic steroids or another immunosuppressive agents (at a dose equivalent of greater than 20 mg prednisone per day) or other immunosuppressive agents)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Reeder, M.D., Study Chair — Mayo Clinic; Thomas E. Witzig, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level -1: Patients receive 5 mg oral everolimus once daily and 5 mg oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 0; Phase II: Dose Level 0: Patients receive 5 mg oral everolimus once daily and 10 mg oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 1: Patients receive 5 mg oral everolimus once daily and 15 mg oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I: Dose Level -1 | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase II: Dose Level 0
Started | 7 | 9 | 9 | 33
Completed | 6 | 9 | 7 | 31
Not Completed | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Treatment Incomplete due to progression | 1 | 0 | 0 | 0
Not completed — Ineligible (miscalculated lab value) | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Fifty-five patients began study treatment and were eligible for response evaluation were pooled and included in this analysis.
Groups:
- All Patients (Everolimus and Lenalidomide): Patients receive oral everolimus once daily and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Patients (Everolimus and Lenalidomide)
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 62 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 54
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Dose-Limiting Toxicity (DLT) (Phase I)
Description: The number of dose-limiting toxic events (DLT) for this combination of drug treatment will determine the Maximum Tolerated Dose (MTD) in subsequent phases of this study. The following events were defined as a DLT: a grade 4+ Neutropenia or platelet count decrease, a grade 4 infection, or any grade 3+ non-hematologic event as assessed using Common Terminology Criteria for Adverse Events (CTCAE) CTEP Version 4.0. Here, the number of patients reporting a DLT are reported
Time Frame: After one 28 day cycle
Population: All Phase 1 patients that began treatment, completed 1 cycle, and were evaluated for cycle 1 toxicity were included in this analysis. Of the 9 registered to Dose Level 1, 2 were ineligible for this endpoint (PD before evaluated and dose error) and 1 cancelled. Phase II patients were not evaluated for dose-limiting toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level -1 | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase II: Dose Level 0
Number analyzed (Participants) | 6 | 9 | 6 | 0
Participants | 1 | 2 | 3 | 0

2. Primary Outcome: Best Response to Dose Level 0
Description: Patients were assessed using the Cheson et al. Revised Response Criteria for Malignant Lymphoma (Cheson, et al 2007). A Complete Response (CR) was defined as the disappearance of all evidence of disease, no palpable nodules and bone marrow cleared on biopsy. A Partial Response (PR) was defined as regression of measureable disease and no new sites, with a 50% decrease in sum of the products of dimension (SPD) of nodal masses, and no increase in spleen or liver size. Patients with Waldenstrom's Macroglobulinemia were eligible to be evaluated as a Minor Response (MR) in which a reduction between 25% and 50% of serum monoclonal IgM was observed. A Progression (PD) was defined as having any new lesions or a 50% increase in the SPD of any previously involved nodes. A Stable Disease (SD) is the absence of any of the previously defined responses.
Time Frame: Up to 5 years
Population: All patients that were registered and treated at Dose Level 0 were pooled and included in this endpoint. 9 patients in Phase I and 32 patients in Phase II were treated and evaluable for this endpoint
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 0: Patients receive 5 mg oral everolimus once daily and 10 mg oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 0
Number analyzed (Participants) | 41
Participants
  Complete Response | 4
  Partial Response | 8
  Minor Response | 1
  Stable Disease | 16
  Progression | 12

3. Secondary Outcome: Overall Survival for All Eligible Patients
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients (Everolimus and Lenalidomide)
Number analyzed (Participants) | 55
months | 20.3 [8.7 to 51.3]

4. Secondary Outcome: Progression-Free Survival For All Eligible Patients
Description: Progression-free survival time is defined as the time from registration to the earliest date of documentation of disease progression. The distribution of progression-free survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients (Everolimus and Lenalidomide)
Number analyzed (Participants) | 55
months | 5.3 [3.0 to 7.0]

5. Secondary Outcome: Duration of Response for All Eligible Patients
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest objective status is first noted to be either a CR or PR to the earliest date progression is documented.
Time Frame: Up to 5 years
Population: All eligible patients that began study treatment and evaluated as a CR, PR or MR during treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients (Everolimus and Lenalidomide)
Number analyzed (Participants) | 15
months | 14.7 [2.8 to 22.0]

6. Secondary Outcome: Time to Treatment Failure for All Eligible Patients
Description: Time to treatment failure is defined to be the time from registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. The distribution of time to treatment failure will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients (Everolimus and Lenalidomide)
Number analyzed (Participants) | 55
months | 4.7 [2.2 to 6.6]

ADVERSE EVENTS:
Description: Adverse Events (AEs) were assessed at the end of every 28 day cycle of treatment. Serious AEs and Other (Not Including Serious) AEs summary tables summarizes AEs assessed for participants who did NOT withdraw from the study (i.e. Withdrawal by Subject in participant flow) and did not have protocol violation (i.e. Protocol Violation in participant flow). All-cause mortality is assessed for participants who did NOT withdraw from the study (i.e. Withdrawal by Subject in participant flow).
Arm/Group | Phase I: Dose Level -1 | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase II: Dose Level 0
All-Cause Mortality (participants affected / at risk) | 6/7 | 6/9 | 7/8 | 18/32
Serious Adverse Events (participants affected / at risk) | 3/7 | 7/9 | 5/7 | 14/32
Other Adverse Events (participants affected / at risk) | 6/7 | 9/9 | 7/7 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level -1 (N=7) | Phase I: Dose Level 0 (N=9) | Phase I: Dose Level 1 (N=7) | Phase II: Dose Level 0 (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 5 (5)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 3 (4)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level -1 (N=7) | Phase I: Dose Level 0 (N=9) | Phase I: Dose Level 1 (N=7) | Phase II: Dose Level 0 (N=32)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (12) | 2 (2) | 8 (27)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 6 (9) | 0 (0) | 17 (61)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 2 (6) | 2 (3) | 6 (15)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (9) | 4 (5) | 17 (39)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (5) | 3 (3) | 9 (12)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 3 (11) | 5 (23) | 2 (2) | 13 (32)
Fatigue (General disorders) | 6 (22) | 7 (38) | 7 (11) | 27 (178)
Fever (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (6) | 10 (32)
Neutrophil count decreased (Investigations) | 3 (12) | 8 (43) | 4 (14) | 25 (159)
Platelet count decreased (Investigations) | 3 (16) | 9 (68) | 5 (15) | 23 (140)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
White blood cell decreased (Investigations) | 4 (18) | 8 (52) | 6 (17) | 26 (137)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (7)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 6 (18) | 5 (7) | 23 (67)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 6 (13) | 2 (3) | 17 (52)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (8) | 2 (2) | 3 (3) | 18 (43)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes